CLINICAL TRIAL: NCT06417463
Title: Role of TIRADS and Bethesda Scoring Systems in Management of Thyroid Nodules
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Keroless Nagy Boles, resident at general surgery department sohag university hospital, Sohag University
Other Study IDs: Soh-Med-24-04-05MS
Record Dates: First submitted 2024-05-12; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: thyroidectomy opeartion — correlation between TIRADS and Bethesda scoring system (preoperative) and final histopathology (postoperative) in cases of thyroidectomy

SUMMARY:
role of TIRADS and Bethesda scoring system in management of thyroid nodules as these methods are ultrasound clasification that helps increase the diagnostic effectiveness of thyroid nodules and reduces the use of preopeative FNA .that nodules are usually divided into diffent categories based on TIRADS and are then referred to FNA and follow up according to variable risk of maligneny.

DETAILED DESCRIPTION:
this study is an observational study will be conducted on patiend with thyroid nodules will be admitted to general surgical department at sohag university hospital . patients will be approved to have single or multinodular goitre and thyroid nodules more than 1 cm . thyroid nodules are very common disease with great clinical importance although most cases are benign and only 4.5% to 6.5% are malignant ... itis necessary to distinguish those cases to reduce frequency of unnecessary thyroidectomies ... ultrasound classification and Fine needle aspiration (FNA) are first line diagnostic procedures and help in decrease cases undergoing unnecessary thyroidectomies as 50% of the nodules removed recently are malignant and the number of patients undergoing surgery is significantly reduced.

ELIGIBILITY:
Inclusion Criteria:

* patients will proved to have single or multinodular goitre thyroid nodules more than 1cm

Exclusion Criteria:

* thyroid nodules less than 1 cm history of thyroid surgery history of radiotherapy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients will proved to have single or multinodular goitre & patients with thyroid nodules more than 1 cm
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-05-12 (Estimated); Primary Completion 2024-10-12 (Estimated); Study Completion 2024-10-12 (Estimated)

PRIMARY OUTCOMES:
managemnt thyroid nodules | 6 months
  correlation between TIRADS and Behtesda scoring systems (preoperative) and final histopathology (post opeartive) in cases of thyroidectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] AlSaedi AH, Almalki DS, ElKady RM. Approach to Thyroid Nodules: Diagnosis and Treatment. Cureus. 2024 Jan 13;16(1):e52232. doi: 10.7759/cureus.52232. eCollection 2024 Jan. PMID 38352091
- [Background] Bojunga J, Trimboli P. Thyroid ultrasound and its ancillary techniques. Rev Endocr Metab Disord. 2024 Feb;25(1):161-173. doi: 10.1007/s11154-023-09841-1. Epub 2023 Nov 10. PMID 37946091
- [Background] Cibas ES, Ali SZ. The 2017 Bethesda System for Reporting Thyroid Cytopathology. Thyroid. 2017 Nov;27(11):1341-1346. doi: 10.1089/thy.2017.0500. PMID 29091573
- [Background] Pemayun TG. Current Diagnosis and Management of Thyroid Nodules. Acta Med Indones. 2016 Jul;48(3):247-257. PMID 27840362